CLINICAL TRIAL: NCT06216418
Title: A Single Center, Prospective, Comparative, Randomized, Double-blinded(Subject, Evaluator), Non-inferiority, Pivotal Clinical Study to Evaluate the Efficacy and Safety of the Polydioxanone Suture 'BRFS-18G-S100WH' Compared to 'MINT Lift FINE+' for Correction of the Nasolabial Folds
Brief Title: Evaluate the Safety and Efficacy of 'BRFS-18G-S100WH' as Compared to 'MINT Lift FINE+' in Subject With Nasolabial Folds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hugel (Industry)
Collaborators: Jworld (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JWD-TH-01
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRFS-18G-S100WH (Experimental)
  Interventions: Device: BRFS-18G-S100WH
- MINT Lift FINE+ (Active Comparator)
  Interventions: Device: MINT Lift FINE+

INTERVENTIONS:
Device: BRFS-18G-S100WH — A facial tissue fixation material made of polydioxanone (PDO).
  Arms: BRFS-18G-S100WH
Device: MINT Lift FINE+ — A facial tissue fixation material made of polydioxanone (PDO).
  Arms: MINT Lift FINE+

SUMMARY:
Evaluate the Safety and Efficacy of 'BRFS-18G-S100WH' as Compared to 'MINT Lift FINE+' in Subject With Nasolabial Folds.

DETAILED DESCRIPTION:
This clinical trial was conducted on patients who wanted to improve both nasolabial folds through facial tissue lifting using facial tissue fixing material 'BRFS-18G-S100WH' made of polydioxanone (PDO). Compared to 'MINT Lift FINE+', we want to confirm whether it has a non-inferior temporary wrinkle improvement effect and can be safely applied to the human body.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age
2. Those who wish to temporarily improve nasolabial folds on both sides of the face and have a score of 3 (Moderate) or 4 (Severe) on the WSRS (Wrinkle Severity Rating Scale)
3. Those who voluntarily decided to participate in this clinical trial and agreed to the subject description and consent form in writing

Exclusion Criteria:

1. A person who has undergone a procedure using filler or facial tissue fixation thread on the facial area.
2. Those who are pregnant or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Improvement rate (%) at 12 weeks after the procedure compared to baseline. | Baseline to week 12
  Improvement rate (%) at 12 weeks after the procedure compared to baseline by an independent evaluator.

SECONDARY OUTCOMES:
WSRS evaluation by an independent evaluator | Baseline to week 4, 8, 24
  Improvement rate (%): 4, 8, and 24 weeks after treatment. Baseline score change (points): 4, 8, 12, and 24 weeks after the procedure.
WSRS evaluation by tester | Baseline to week 4, 8, 24
  Improvement rate (%): 4, 8, and 24 weeks after treatment. Baseline score change (points): 4, 8, 12, and 24 weeks after the procedure.
Satisfaction level (%) at 4, 8, 12, and 24 weeks after the procedure compared to the baseline. | Baseline to week 4, 8, 12, 24
  Satisfaction level (%) at 4, 8, 12, and 24 weeks after the procedure compared to the baseline by the subject

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel Inc., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No